CLINICAL TRIAL: NCT07359040
Title: Mechanisms of Enhanced Efficacy of Ivonescimab in Neoadjuvant Therapy for Non-Small Cell Lung Cancer
Brief Title: Mechanism of Enhanced Efficacy of Ivonescimab in Neoadjuvant Therapy for Non-Small Cell Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Fan, MD, Vice President, Peking University People's Hospital
Other Study IDs: BRWEP2024W034080205
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Neoadjuvant Therapy; PD-1 Inhibitors; Immunotherapy
Keywords: Neoajuvant therapy; Ivonescimab; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ivonescimab neoadjuvant therapy group: Patients in this group will receive ivonescimab as neoadjuvant therapy
  Interventions: Drug: Ivonescimab
- PD-1 inhibitors neoadjuvant therapy group: Patients in this group will receive other PD-1 inhibitors as neoadjuvant therapy
  Interventions: Drug: PD-1 Inhibitors

INTERVENTIONS:
Drug: Ivonescimab — Patients in the experimental group will receive ivonescimab as neoadjuvant therapy.
  Groups: Ivonescimab neoadjuvant therapy group
Drug: PD-1 Inhibitors — Patients in the positive control group will receive PD-1 inhibitors monotherapy as neoadjuvant treatment.
  Groups: PD-1 inhibitors neoadjuvant therapy group

SUMMARY:
This study primarily aims to compare the efficacy and safety of Ivonescimab (a PD-1/VEGF bispecific antibody) with conventional PD-1 inhibitors in the neoadjuvant treatment of non-small cell lung cancer, as well as to explore the potential mechanisms underlying its enhanced therapeutic effects, thereby providing experimental data to support the clinical application of Ivonescimab.

DETAILED DESCRIPTION:
Lung cancer is one of the leading causes of cancer-related deaths in China and worldwide, imposing a significant societal burden. Although comprehensive treatment strategies centered around surgery have improved patient prognosis, and perioperative immunotherapy has profoundly reshaped the therapeutic landscape, this field still faces substantial knowledge gaps and key challenges.

This study focuses on Ivonescimab, a first-in-class PD-1/VEGF bispecific antibody. Ivonescimab simultaneously blocks PD-1 to reactivate antitumor immune response by releasing T-cell inhibition and inhibits VEGF to suppress tumor angiogenesis while modulating the immunosuppressive tumor microenvironment. The primary objectives of this research are to evaluate the efficacy and safety of Ivonescimab compared with conventional immunotherapy and to investigate its potential mechanisms of action, thereby providing scientific evidence to support its clinical application.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-small cell lung cancer (Stage IB-IIIB) who require radical surgery following neoadjuvant therapy.

Exclusion Criteria:

1. Histology of other malignant tumors, including concurrent malignant tumors of other organ systems;
2. Unresectable advanced disease (Stage IV) or locally advanced unresectable (Stage IIIC);
3. Pregnancy or lactation;
4. Insufficient sample quality;
5. Severe organ dysfunction (e.g. cardiac or renal insufficiency);
6. Other judgments by the Investigator that the patient should not participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study primarily involves patients with small cell lung cancer who require neoadjuvant immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-12-21 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR | At surgery (typically 3-6 months post-treatment initiation)
  Pathologic Complete Response (pCR) is defined as the absence of residual tumor in both the primary lung tumor site and all sampled regional lymph nodes after neoadjuvant immunotherapy, confirmed through systematic pathological examination of the surgical specimen.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | At surgery (typically 3-6 months post-treatment initiation)
  Major Pathologic Response (MPR) is defined as the presence of ≤10% residual viable tumor cells in both the primary lung tumor site and sampled regional lymph nodes after neoadjuvant immunotherapy, confirmed through systematic pathological examination of the surgical specimen.
Objective Response Rate (ORR) | After two cycles or four cycles of neoadjuvant therapy (each cycle is 21 days).
  ORR is defined as the proportion of patients achieving either a complete response (CR; disappearance of all target lesions) or partial response (PR; ≥30% reduction in the sum of target lesion diameters) during or after neoadjuvant immunotherapy, as assessed by serial imaging (CT/PET-CT) using iRECIST criteria.
Event-free Survival (EFS) | Through study completion, an average of 2 years.
  Time from randomization to the occurrence of any of the following events: disease progression, recurrence, discontinuation of treatment due to toxicity, initiation of new anticancer therapy, or death from any cause.
Overall Survival (OS) | Through study completion, an average of 2 years.
  Time from randomization to death from any cause.
MRD (minimal residual disease) dynamics after neoadjuvant immunotherapy | Periprocedural and every three to six months post-treatment (up to three years).
  Postoperative dynamics of ctDNA-based MRD and timely detection of recurrence or metastasis in lung cancer patients receiving neoadjuvant immunotherapy.
Immune-Related Adverse Event (irAE) Incidence | Periprocedural and up to 6 months post-treatment.
  Frequency and severity of adverse events (e.g., rash, colitis) related to immunotherapy, graded using standardized criteria like CTCAE (Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wang L, Luo Y, Ren S, Zhang Z, Xiong A, Su C, Zhou J, Yu X, Hu Y, Zhang X, Dong X, Meng S, Wu F, Hou X, Dai Y, Song W, Li B, Wang ZM, Xia Y, Zhou C. A Phase 1b Study of Ivonescimab, a Programmed Cell Death Protein-1 and Vascular Endothelial Growth Factor Bispecific Antibody, as First- or Second-Line Therapy for Advanced or Metastatic Immunotherapy-Naive NSCLC. J Thorac Oncol. 2024 Mar;19(3):465-475. doi: 10.1016/j.jtho.2023.10.014. Epub 2023 Oct 23. PMID 37879536
- [Result] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- [Result] Zhao S, Zhao H, Yang W, Zhang L. The next generation of immunotherapies for lung cancers. Nat Rev Clin Oncol. 2025 Aug;22(8):592-616. doi: 10.1038/s41571-025-01035-9. Epub 2025 Jun 17. PMID 40528044
- [Result] Chen Z, Yang F, Jiang Z, Sun L, Wu L, Han Z, Fan Y, Zhao Y, Li X, Xu H, Meng X, Liu Y, Zhang Z, Luo H, Ma X, Ma X, Shi Q, Zhang Z, Yang R, Wang P, Pan P, Ai X, Li J, Pu X, Wang Z, Fang J, He M, He Y, Guo S, Li J, Wang H, Zhang J, Chu Q, Liu X, Ying S, Wu H, Sun H, Ji Y, Zhou M, Cao C, Tang K, Li Z, Li D, Zhang Z, Li J, Zhou J, Yang H, Du Y, Yang H, Shi J, Chen H, Li W, Lu D, Hu M, Maxwell Wang Z, Li B, Xia M, Lu S. Ivonescimab plus chemotherapy versus tislelizumab plus chemotherapy as first-line treatment for advanced squamous non-small-cell lung cancer (HARMONi-6): a randomised, double-blind, phase 3 trial. Lancet. 2025 Nov 1;406(10515):2078-2088. doi: 10.1016/S0140-6736(25)01848-3. Epub 2025 Oct 19. PMID 41125109
- [Result] Xiong A, Wang L, Chen J, Wu L, Liu B, Yao J, Zhong H, Li J, Cheng Y, Sun Y, Ge H, Yao J, Shi Q, Zhou M, Chen B, Han Z, Wang J, Bu Q, Zhao Y, Chen J, Nie L, Li G, Li X, Yu X, Ji Y, Sun D, Ai X, Chu Q, Lin Y, Hao J, Huang D, Zhou C, Shan J, Yang H, Liu X, Wang J, Shang Y, Mei X, Yang J, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhou C. Ivonescimab versus pembrolizumab for PD-L1-positive non-small cell lung cancer (HARMONi-2): a randomised, double-blind, phase 3 study in China. Lancet. 2025 Mar 8;405(10481):839-849. doi: 10.1016/S0140-6736(24)02722-3. PMID 40057343